CLINICAL TRIAL: NCT06833047
Title: Does Boredom Affect Mechanical Pain Thresholds
Acronym: BEAMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Helena Gunnarsson, Dr, Linnaeus University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Dnr 2024-07849-01
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Pain Threshold; Healthy
Keywords: Pain Thresholds; Pain; Boredom
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to different conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Boredom (Experimental): The participant will watch a short video with boring content.
  Interventions: Behavioral: Emotional intervention
- Distraction control (Experimental): The participant will watch a short video with positively valenced content.
  Interventions: Behavioral: Emotional intervention
- Control (No Intervention): The participant will wait for 2.30 minutes without any instructions of what to think about.

INTERVENTIONS:
Behavioral: Emotional intervention — Participants will receive different emotional interventions such as boredom, positive valence, mind-wandering.
  Arms: Boredom; Distraction control

SUMMARY:
The purpose of this study is to investigate if the feeling of boredom could influence mechanical pain thresholds.

DETAILED DESCRIPTION:
Participants will be randomized into 3 different groups watching different short video-clips (2.30 min). The boredom group will watch a boring video about ploughing, the distraction control group will watch a positively valenced video, the control group will just wait for 2.30 min, without any instructions about what to think about. Pressure pain thresholds will be measured with an algometer before and after the video-clip interventions.

ELIGIBILITY:
Inclusion Criteria:

* No pain at the test session
* Swedish fluency.

Exclusion Criteria:

* Pain anywhere in the body during the test session
* known neurological disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Pressure pain thresholds | 30 minutes
  Pressure Pain thresholds will be measured over the right and left m. trapezius and over the right and left m. tibialis anterior.

CONTACTS AND LOCATIONS:
Locations (1):
- Linnaeus University, Vaxjo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The anonymous data collected will be shared. Any information that could possibly be used to identify a participant (education) will be removed.